CLINICAL TRIAL: NCT01658579
Title: A 16-week, Randomized, Open-label, Controlled Study Comparing the Efficacy and Safety of a New Formulation of Insulin Glargine Versus Lantus in Patients With Type 1 Diabetes Mellitus
Brief Title: Comparison of a New Formulation of Insulin Glargine With Lantus in Patients With Type 1 Diabetes Mellitus on Basal Plus Mealtime Insulin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PDY12777; U1111-1130-3593 (Other: UTN)
Record Dates: First submitted 2012-07-26; First posted 2012-08-07 (Estimated); Results first posted 2015-05-07 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- HOE901-U300 Morning Then Evening (Experimental): HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily in morning for 8 weeks during treatment period A, followed by once daily in evening for 8 weeks during treatment period B. Dose titration seeking fasting plasma glucose 4.4-7.2 millimole per liter (mmol/L).
  Interventions: Drug: HOE901-U300 (new formulation of insulin glargine)
- HOE901-U300 Evening Then Morning (Experimental): HOE901-U300 (new insulin glargine 300 U/mL) SC injection once daily in evening for 8 weeks during treatment period A, followed by once daily in morning for 8 weeks during treatment period B. Dose titration seeking fasting plasma glucose 4.4-7.2 mmol/L.
  Interventions: Drug: HOE901-U300 (new formulation of insulin glargine)
- Lantus Morning Then Evening (Active Comparator): Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily in morning for 8 weeks during treatment period A, followed by once daily in evening for 8 weeks during treatment period B. Dose titration seeking fasting plasma glucose 4.4-7.2 mmol/L.
  Interventions: Drug: Lantus (insulin glargine)
- Lantus Evening Then Morning (Active Comparator): Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily in evening for 8 weeks during treatment period A, followed by once daily in morning for 8 weeks during treatment period B. Dose titration seeking fasting plasma glucose 4.4-7.2 mmol/L.
  Interventions: Drug: Lantus (insulin glargine)

INTERVENTIONS:
Drug: HOE901-U300 (new formulation of insulin glargine)
  Arms: HOE901-U300 Evening Then Morning; HOE901-U300 Morning Then Evening
Drug: Lantus (insulin glargine)
  Arms: Lantus Evening Then Morning; Lantus Morning Then Evening

SUMMARY:
Primary Objective:

* To compare the glucose control during treatment with a new formulation of insulin glargine and Lantus in adult participants with type 1 diabetes mellitus

Secondary Objectives:

* To compare a new formulation of insulin glargine and Lantus given in the morning or in the evening
* To compare the incidence and frequency of hypoglycemic episodes
* To assess the safety and tolerability of the new formulation of insulin glargine

DETAILED DESCRIPTION:
* Up to 4-week screening period;
* 16-week open-label comparative efficacy and safety treatment period;
* 4-week post-treatment safety follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Participants with Type 1 diabetes mellitus

Exclusion criteria:

* HbA1c greater than (>) 9% (at screening)
* Participants receiving >0.5 U/kg body weight basal insulin in the last 30 days prior to screening visit
* Participants not on stable insulin dose (+/- 20% total basal insulin dose) in the last 30 days prior to screening visit
* Less than 1 year on any basal plus mealtime insulin
* Participants using pre-mix insulins, human regular insulin as mealtime insulin and/or any antidiabetic drugs other than basal insulin and mealtime analogue insulin in the last 3 months before screening visit
* Use of an insulin pump in the last 6 months before screening visit;
* Any contraindication to use of insulin glargine as defined in the national product label
* Not willing to inject insulin glargine as assigned by the randomization process once daily in the morning or evening
* Hospitalization for diabetic ketoacidosis or history of severe hypoglycemia (requiring 3rd party assistance) in the last 6 months prior to randomization
* Initiation of any glucose-lowering agents in the last 3 months before screening visit
* Weight change of greater than equal to (>=) 5 kg during the last 3 months prior to screening visit
* Unstable proliferative diabetic retinopathy or any other rapidly progressive diabetic retinopathy or macular edema likely to require laser, surgical treatment or injectable drugs during the study period

The above information is not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (3):
- United States (3):
  - Investigational Site Number 840002, Temecula, California
  - Investigational Site Number 840001, Minneapolis, Minnesota
  - Investigational Site Number 840003, Portland, Oregon

REFERENCES:
- [Derived] Bergenstal RM, Bailey TS, Rodbard D, Ziemen M, Guo H, Muehlen-Bartmer I, Ahmann AJ. Comparison of Insulin Glargine 300 Units/mL and 100 Units/mL in Adults With Type 1 Diabetes: Continuous Glucose Monitoring Profiles and Variability Using Morning or Evening Injections. Diabetes Care. 2017 Apr;40(4):554-560. doi: 10.2337/dc16-0684. Epub 2017 Jan 23. PMID 28115474

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 85 participants were screened, of whom 26 participants were screen failures and 59 participants were randomized. The data for outcome measures was planned to be reported for combined reporting arms (HOE901-U300 Combined and Lantus Combined).
Groups:
- HOE901-U300 Morning Then Evening: HOE901-U300 (new insulin glargine 300 units per milliliter [U/mL]) subcutaneous (SC) injection once daily in morning for 8 weeks during treatment period A, followed by once daily in evening for 8 weeks during treatment period B. Dose titration seeking fasting plasma glucose 4.4-7.2 millimole per liter (mmol/L) (80-130 milligram per deciliter [mg/dL]).
- HOE901-U300 Evening Then Morning: HOE901-U300 SC injection once daily in evening for 8 weeks during treatment period A, followed by once daily in morning for 8 weeks during treatment period B. Dose titration seeking fasting plasma glucose 4.4-7.2 mmol/L (80-130 mg/dL).
- Lantus Morning Then Evening: Lantus (HOE901-U100, insulin glargine 100 U/mL) SC injection once daily in morning for 8 weeks during treatment period A, followed by once daily in evening for 8 weeks during treatment period B. Dose titration seeking fasting plasma glucose 4.4-7.2 mmol/L (80-130 mg/dL).
- Lantus Evening Then Morning: Lantus SC injection once daily in evening for 8 weeks during treatment period A, followed by once daily in morning for 8 weeks during treatment period B. Dose titration seeking fasting plasma glucose 4.4-7.2 mmol/L (80-130 mg/dL).
Period: Treatment Period A
Arm/Group | HOE901-U300 Morning Then Evening | HOE901-U300 Evening Then Morning | Lantus Morning Then Evening | Lantus Evening Then Morning
Started | 15 | 15 | 15 | 14
Completed | 14 | 15 | 14 | 13
Not Completed | 1 | 0 | 1 | 1
Not completed — Other | 0 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0 | 0
Period: Treatment Period B
Arm/Group | HOE901-U300 Morning Then Evening | HOE901-U300 Evening Then Morning | Lantus Morning Then Evening | Lantus Evening Then Morning
Started | 14 | 15 | 14 | 13
Completed | 14 | 15 | 14 | 12
Not Completed | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Randomized population: all screened participants (who originally met inclusion criteria and signed informed consent) allocated to a treatment arm and recorded in Interactive Voice/Web Response System (IVRS/IWRS) database, regardless of whether treatment was used or not. Participants were analyzed in treatment arm to which they were randomized.
Groups:
- HOE901-U300 Morning Then Evening: HOE901-U300 SC injection once daily in morning for 8 weeks during treatment period A, followed by once daily in evening for 8 weeks during treatment period B.
- HOE901-U300 Evening Then Morning: HOE901-U300 SC injection once daily in evening for 8 weeks during treatment period A, followed by once daily in morning for 8 weeks during treatment period B.
- Lantus Morning Then Evening: Lantus SC injection once daily in morning for 8 weeks during treatment period A, followed by once daily in evening for 8 weeks during treatment period B.
- Lantus Evening Then Morning: Lantus SC injection once daily in evening for 8 weeks during treatment period A, followed by once daily in morning for 8 weeks during treatment period B.
- Total: Total of all reporting groups
Arm/Group | HOE901-U300 Morning Then Evening | HOE901-U300 Evening Then Morning | Lantus Morning Then Evening | Lantus Evening Then Morning | Total
Number analyzed (Participants) | 15 | 15 | 15 | 14 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.6 (14.6) | 46.2 (15.9) | 39.7 (12.5) | 47.6 (14.1) | 44.2 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 2 | 4 | 10 | 27
  Male | 4 | 13 | 11 | 4 | 32
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 27.5 (4.9) | 27.4 (5.0) | 28.3 (6.2) | 26.1 (5.1) | 27.3 (5.3)
Glycated Hemoglobin (HbA1c) [Number; unit: participants]
  Less Than (<) 8 | 11 | 14 | 12 | 12 | 49
  Greater Than or Equal to (>=) 8 | 4 | 1 | 3 | 2 | 10
Duration of Diabetes [Median (Full Range); unit: years] | 16.8 [3 to 48] | 23.9 [2 to 54] | 20.6 [5 to 47] | 16.7 [6 to 44] | 20.7 [2 to 54]
Basal Insulin Daily Dose [Mean (Standard Deviation); unit: units per kilogram (U/kg)] — Number of participants analyzed for this baseline characteristics =15, 14, 15, and 13 for each reporting group, respectively.
  units per kilogram (U/kg) | 0.309 (0.086) | 0.283 (0.088) | 0.341 (0.100) | 0.267 (0.055) | 0.301 (0.087)
Total Insulin Daily Dose [Mean (Standard Deviation); unit: U/kg] — Number of participants analyzed for this baseline characteristics = 13, 13, 13, 13 for each reporting group, respectively.
  U/kg | 0.600 (0.237) | 0.620 (0.179) | 0.677 (0.204) | 0.513 (0.115) | 0.603 (0.193)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time in Target Plasma Glucose Range (4.4-7.8 mmol/L [80-140 mg/dL])
Description: Percentage of time with glucose within glycemic range (4.4-7.8 mmol/L) was assessed by the total time within glycemic range divided by the length of the assessment interval.
Time Frame: Up to Week 16 (assessed at Weeks 7-8 in Period A and Weeks 15-16 in Period B)
Population: Continuous glucose monitoring (CGM) population: All participants who received at least 1 dose, had evaluable post-baseline CGM data, irrespective of compliance. Number of participants analyzed = participants with baseline, Weeks 7-8 (Period A) and/or Weeks 15-16 (Period B) CGM assessment. Missing data imputed using last observation carried forward.
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Groups:
- HOE901-U300 Combined: HOE901-U300 SC injection once daily in morning or evening for 8 weeks during treatment period A, followed by once daily in evening or morning for 8 weeks during treatment period B.
- Lantus Combined: Lantus SC injection once daily in morning or evening for 8 weeks during treatment period A, followed by once daily in evening or morning for 8 weeks during treatment period B.
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 30 | 27
percentage of time | 31.75 (1.5) | 30.99 (1.58)
Statistical Analysis 1: Comparison: HOE901-U300 Combined vs Lantus Combined; Analysis was performed using a linear mixed model with treatment and period as fixed effects, and participant as random effect; Test type: Superiority or Other; p = 0.7304, Linear Mixed Model; Least Squares (LS) Mean Difference = 0.75, 95% CI 2-sided [-3.614 to 5.124], Standard Error of Mean 2.179

2. Secondary Outcome: Percentage of Time Above the Upper Limit of Glycemic Range (Greater Than [>] 7.8 mmol/L [(140 mg/dL])
Description: Percentage of time with glucose above the upper limit of glycemic range (>7.8 mmol/L) was assessed by the total time above the upper limit of glycemic range divided by the length of the assessment interval.
Time Frame: Up to Week 16 (assessed at Weeks 7-8 in Period A and Weeks 15-16 in Period B)
Population: CGM population. Number of participants analyzed = participants with baseline, Weeks 7, 8 (Period A), and/or Weeks 15, 16 (Period B) CGM assessment. Missing data imputed using last observation carried forward (LOCF).
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 30 | 27
percentage of time | 58.24 (2.09) | 57.38 (2.2)

3. Secondary Outcome: Percentage of Time Below The Lower Limit of Glycemic Range (<4.4 mmol/L [80 mg/dL])
Description: Percentage of time with glucose below the lower limit of glycemic range (<4.4 mmol/L) was assessed by the total time below the lower limit of glycemic range divided by the length of the assessment interval.
Time Frame: Up to Week 16 (assessed at Weeks 7-8 in Period A and Weeks 15-16 in Period B)
Population: CGM population. Number of participants analyzed = participants with baseline, Weeks 7, 8 (Period A), and/or Weeks 15, 16 (Period B) CGM assessment. Missing data imputed using LOCF.
Measure: Least Squares Mean (Standard Error); unit: percentage of time
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 30 | 27
percentage of time | 10.01 (1.02) | 11.64 (1.08)

4. Secondary Outcome: Evaluation of Diurnal Glucose Exposure, Variability, and Stability
Description: The diurnal glucose exposure is measured as the average diurnal glucose concentration, diurnal glucose variability is measured by interquartile range (IQR), that is, average distance between the 25th and the 75th point-wise percentiles and diurnal glucose stability is assessed in terms of the mean absolute rate of change (mmol/l), that is, the area under the absolute rate of change of the median curve (based on the median point values between two adjacent hourly basket intervals), divided by the length of the assessment interval.
Time Frame: Up to Week 16 (assessed at Weeks 7-8 in Period A and Weeks 15-16 in Period B)
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 30 | 27
mmol/L
  Diurnal Glucose Exposure | 8.869 (0.24) | 8.910 (0.26)
  Diurnal Glucose Stability | 0.673 (0.03) | 0.703 (0.03)
  Diurnal Glucose Variability | 4.931 (0.22) | 5.279 (0.23)

5. Secondary Outcome: Percentage of Time in Target Plasma Glucose Range (4.4-7.8 mmol/L [80-140 mg/dL]) in the Last Four Hours of Each Dosing Interval at Weeks 7 and 8 in Period A and Weeks 15 and 16 in Period B
Description: as for outcome 1
Time Frame: Weeks 7-8 in Period A and Weeks 15-16 in Period B
Population: CGM population. Number of participants analyzed = participants with baseline, Weeks 7, 8 (Period A), and/or Weeks 15, 16 (Period B) CGM assessment, and n = participants with assessment at specified time-point.
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 29 | 27
percentage of time
  Week 7, 8 (n=28, 27) | 32.08 (14.74) | 29.07 (13.82)
  Week 15, 16 (n=29, 26) | 33.02 (13.48) | 28.70 (14.57)

6. Secondary Outcome: Change in HbA1c From Baseline to Week 8 and 16
Time Frame: Baseline, Week 8, 16
Population: Modified Intent-to-Treat population: randomized participants who received at least 1 dose; had baseline, at least 1 post-baseline efficacy assessment; irrespective of compliance. Number of participants analyzed = participants with baseline, Week 8 and/or 16 HbA1c assessment, n = participants with HbA1c assessment at specified time. LOCF applied.
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 29 | 27
percentage of hemoglobin
  Week 8 (n= 29, 20) | -0.22 (0.48) | -0.23 (0.54)
  Week 16 (n= 28, 27) | -0.44 (0.51) | -0.22 (0.58)

7. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 8 and 16
Time Frame: Baseline, Week 8, 16
Population: Modified Intent-to-Treat population. Number of participants analyzed = participants with baseline, Week 8 and/or 16 FPG assessment, n = participants with FPG assessment at specified time. Missing data imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 24 | 23
mmol/L
  Week 8 (n=24, 23) | -0.89 (5.04) | -0.10 (5.81)
  Week 16 (n= 24, 22) | -0.99 (5.27) | 0.78 (4.92)

8. Secondary Outcome: Change in Average 7-Point Self-Monitored Plasma Glucose (SMPG) Profile From Baseline to Week 8 and 16
Description: Change in average of 7-point SMPG. 7-point SMPG was assessed starting with a measurement at before breakfast and 2 hours after breakfast; before and 2 hours after lunch; before and 2 hours after dinner; at bedtime.
Time Frame: Baseline, Week 8, 16
Population: Modified Intent-to-Treat population. Number of participants analyzed = participants with baseline, Week 8 and/or 16 7-point SMPG assessment, n = participants with 7-point SMPG assessment at specified time. Missing data imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 22 | 22
mmol/L
  Week 8 | -0.39 (1.84) | 0.39 (1.54)
  Week 16 | -0.47 (1.31) | 0.58 (2.13)

9. Secondary Outcome: Change in Basal Insulin Daily Dose From Baseline to Week 8 and 16
Time Frame: Baseline, Week 8, 16
Population: Modified Intent-to-Treat population. Here n = participants with basal insulin dose assessment at specified time-point. Missing data imputed using LOCF.
Measure: Mean (Standard Deviation); unit: U/kg
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 30 | 29
U/kg
  Week 8 (n= 30, 29) | 0.06 (0.09) | 0.03 (0.09)
  Week 16 (n=29, 27) | 0.05 (0.09) | 0.03 (0.08)

10. Secondary Outcome: Percentage of Participants With Hypoglycemia (All and Nocturnal) Events From Baseline Up to Week 16
Description: Hypoglycemia events were Severe hypoglycemia (an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions); Documented symptomatic hypoglycemia (typical symptoms of hypoglycemia with plasma glucose level of <=3.9 mmol/L [70 mg/dL]); Asymptomatic hypoglycemia (no typical symptoms of hypoglycemia but plasma glucose level <=3.9 mmol/L); Probable symptomatic hypoglycemia (an event during which symptoms of hypoglycemia were not accompanied by a plasma glucose determination, but was presumably caused by a plasma glucose level <=3.9 mmol/L, symptoms treated with oral carbohydrate without a test of plasma glucose); Relative hypoglycemia (an event during which the person with diabetes reported any of the typical symptoms of hypoglycemia, and interpreted the symptoms as indicative of hypoglycemia, but plasma glucose level >3.9 mmol/L); Severe and/or confirmed a hypoglycemia (plasma glucose <=3.9 mmol/L).
Time Frame: Up to Week 16
Population: Safety population: all randomized participants who were exposed to at least one dose, regardless of amount of treatment administered. In the event of participants having received treatments different from those assigned according to the randomization schedule, safety analyses were conducted according to treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 Combined | Lantus Combined
Number analyzed (Participants) | 30 | 29
percentage of participants
  Any Hypoglycemia Event: All Hypoglycemia | 100 | 100
  Severe Hypoglycemia: All Hypoglycemia | 3.3 | 10.3
  Documented Symptomatic: All Hypoglycemia | 93.3 | 96.6
  Asymptomatic: All Hypoglycemia | 86.7 | 96.6
  Probable Symptomatic: All Hypoglycemia | 16.7 | 27.6
  Relative: All Hypoglycemia | 0.0 | 6.9
  Severe and/or Confirmed: All Hypoglycemia | 100 | 100
  Any Hypoglycemia Event: Nocturnal Hypoglycemia | 80.0 | 93.1
  Severe Hypoglycemia: Nocturnal Hypoglycemia | 0.0 | 6.9
  Documented Symptomatic: Nocturnal Hypoglycemia | 66.7 | 79.3
  Asymptomatic: Nocturnal Hypoglycemia | 40.0 | 48.3
  Probable Symptomatic: Nocturnal Hypoglycemia | 3.3 | 10.3
  Relative: Nocturnal Hypoglycemia | 0.0 | 6.9
  Severe and/or Confirmed: Nocturnal Hypoglycemia | 80.0 | 93.1

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Week 16) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the 'on treatment period' (the time from first dose of study drug up to 2 days after the last dose of study drug). Analysis was done on safety population.
Arm/Group | HOE901-U300 Combined | Lantus Combined
Serious Adverse Events (participants affected / at risk) | 1/30 | 0/29
Other Adverse Events (participants affected / at risk) | 18/30 | 17/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 Combined (N=30) | Lantus Combined (N=29)
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 Combined (N=30) | Lantus Combined (N=29)
Nasopharyngitis (Infections and infestations) | 9 | 6
Influenza (Infections and infestations) | 2 | 3
Headache (Nervous system disorders) | 2 | 4
Migraine (Nervous system disorders) | 2 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Nausea (Gastrointestinal disorders) | 2 | 1
Vomiting (Gastrointestinal disorders) | 0 | 3
Implant site bruising (General disorders) | 3 | 0
Pyrexia (General disorders) | 3 | 2
Fatigue (General disorders) | 2 | 2
Weight increased (Investigations) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.